CLINICAL TRIAL: NCT04734977
Title: Clinical Effectiveness of High-Intensity Laser Therapy in Patients With Cervical Radiculopathy: A Randomized Study of Double Blınd With Sham Control
Brief Title: Clinical Effectiveness of High-Intensity Laser Therapy in Patients With Cervical Radiculopathy:
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Afyonkarahisar Health Sciences University (Other)
Responsible Party: Principal Investigator, Songül İnce, Research Assistant Doctor, Afyonkarahisar Health Sciences University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NEHILT2021
Record Dates: First submitted 2021-01-25; First posted 2021-02-02 (Actual); Last update posted 2022-09-23 (Actual); Status verified 2022-09

CONDITIONS: Radiculopathy; Musculoskeletal Diseases; Cervical Pain; Cervical Radicular Pain; Cervical Disc Disease
Keywords: High Intensity Laser Therapy; Cervical Radicular Pain; Radiculopathy
MeSH Terms: conditions — Radiculopathy; Musculoskeletal Diseases; Neck Pain | interventions — Exercise Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- HILT+exercise (Experimental): Patients received pulsed laser treatment, using a HIRO 3 device (ASA Laser, Arcugnano, Italy), five times a week for a period of four weeks, and one session per day for a total of 20 sessions. A 3-phase treatment program was performed in each session, and the patients were then given a daily exercise program once a day by a physiotherapist.
  Interventions: Device: High-intensity laser therapy (HILT); Other: Therapeutic Exercise
- Sham HILT+exercise (Sham Comparator): Sham therapy was applied in five sessions a week for four weeks, with a total of 20 sessions a day, with no current flowing through the device. This was followed by the exercise programs described above, performed once a day with the physiotherapist.
  Interventions: Device: Sham high-intensity laser therapy (Sham HILT); Other: Therapeutic Exercise
- Exercise only (Active Comparator): Exercise program was applied in five sessions a week for four weeks, with a total of 20 sessions a day.
  Interventions: Other: Therapeutic Exercise

INTERVENTIONS:
Device: High-intensity laser therapy (HILT) — High intensity laser therapy-Patients received pulsed laser treatment, using a HIRO 3 device (ASA Laser, Arcugnano, Italy), five times a week for a period of four weeks, and one session per day for a total of 20 sessions. A 3-phase treatment program was performed in each session.
  Arms: HILT+exercise
Device: Sham high-intensity laser therapy (Sham HILT) — Sham High intensity laser therapy was applied in five sessions a week for four weeks, with a total of 20 sessions a day, with no current flowing through the device using a HIRO 3 device (ASA Laser, Arcugnano, Italy).
  Arms: Sham HILT+exercise
Other: Therapeutic Exercise — As therapeutic exercise program; active cervical ROM, cervical isometric and progressive (self-exercise with Thera-Band) strengthening muscles; trapezius, scalene, rhomboid, levator scapular, pectoral, suboccipital muscles stretching exercises, scapular stabilization exercises.It was planned to implement a total of 20 sessions 5 days a week for 4 weeks, for approximately 30 minutes.
  Exercises will be performed by a trained (at least 5 years experienced) physiotherapist, three times a day, in 3 sets, 10 repetitions.

SUMMARY:
This investigation aims to investigate the effect of high intensity laser therapy on radicular symptoms, neuropathic pain, cervical range of motion and quality of life in patients with cervical radiculopathy compared to cervical therapeutic exercises.

DETAILED DESCRIPTION:
Most cases of cervical radiculopathy are due to cervical spondylosis or disc herniation. As the age progresses, disintegration of the disc causes a decrease in disc height and foraminal narrowing. The decreased disc height then results in hypertrophy due to vertebral loading in the intervertebral joints of Luschka. This leads to foraminal stenosis and cervical radiculopathy.If cervical radiculopathy is due to disc herniation, its mechanism is explained by the impact of the nerve root with the disc material and causing nerve damage by both mechanical and chemical effects.Non-operative treatment of cervical radiculopathy consists of a number of different modalities including immobilization, physical therapy, traction, manipulation,drug therapy, cervical steroid injection and laser therapy.The physiological effects of high intensity laser therapy(HILT) reduce the release of histamine and bradykinin from inflammatory tissue and increase the pain threshold. In addition, laser light reduces the secretion of substance P from peripheral nociceptors, thereby reducing the perception of pain and preventing the development of hyperalgesia. The laser analgesic effect is due to the increased secretion of endogenous opioids such as β-endorphins, where pain is centrally inhibited.

This investigation was designed double-blind prospective sham controlled randomized study. Participants were randomized into 3 groups: HILT + therapeutic exercise, sham HILT + therapeutic exercise, and only therapeutic exercise.

As evaluation parameters, cervical range of motion, Visual Pain Scale (VAS) Neck, Visual Pain Scale (VAS) Arm, SF (Short form) -36 Quality of Life Scale, Pain Detect Pain questionnaire, Cervical Radiculopathy Impact Scale ) will be evaluated with.It was planned that the evaluations were made and recorded by a blinded physician to the groups at the beginning of the treatment, at the end of the treatment and at the 3rd month controls.

.

ELIGIBILITY:
Inclusion Criteria: Eligible patients aged 20-65 years old with pain in the cervical spine and arm pain with or without neck pain lasting for at least one month. Patients were included in the study

1. radicular clinical symptoms
2. cervical disc herniation and degenerative changes diagnosed with cervical MR
3. radiculopathy findings on Electromyography (EMG) and Nerve Conduction Studies

Exclusion Criteria:

1. Pregnancy
2. Inflammatory rheumatologic diseases
3. Malignity
4. Structural deformity
5. Previous surgery related to the cervical spine
6. Cervical spinal stenosis
7. Lokal corticosteroid injections
8. Medications for neuropathic pain such as pregabalin or gabapentin
9. Carpal tunnel syndrome, cubital tunnel syndrome
10. Shoulder pathology

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2022-09-22 (Actual); Study Completion 2022-09-22 (Actual)

PRIMARY OUTCOMES:
Change from baseline visual analog scale (VAS) neck and arm pain at 4th and 12th week | up to 12th week
  Pain intensity was measured with visual analogue scale for pain (0-10 mm; 0 means no pain, 10 means severe pain) which is used to measure musculoskeletal pain with very good reliability and validity.

SECONDARY OUTCOMES:
Change from baseline quality of life (short form 36 (SF-36)) at 4th and 12th weeks | up to 12th week
  This is a self-administered scale, which is widely used to measure the quality of life. It was developed to measure the quality of life in patients who have physical illnesses; however, it can also be successfully used in healthy individuals and patients who have psychiatric diseases. SF-36 includes 36 items and surveys eight domains of health, such as physical functionality, physical role limitations, pain, general health, vitality, social functionality, emotional role limitations, and mental health. Total score was between 0 ( disability) and 100 (no disability). Every subgroup of the questionnaire has a score scale between 0 and 100. Every increase in the subgroup of SF-36 questionnaire, which is a positive scoring system, indicates increase in quality of life related to health.
Change from baseline range of motion of cervical spine measurements with goniometer at 4th and 12th weeks | up to 12th week
  cervical flexion, extension ,lateral flexion ,rotations(goniometric measurement results in units of degrees)
Change from baseline Neck Dısabılıty Index (NDI) at 4th and 12th weeks | up to 12th week
  The Neck Disability Index (NDI) is designed to measure neck-specific disability. The questionnaire has 10 items concerning pain and activities of daily living including personal care, lifting, reading, headaches, concentration, work status, driving, sleeping and recreation. Each question measures from 0 to 5, the total score out of 100 is calculated.
Change from baseline Cervical Radiculopathy Impact Scale(CRIS) at 4th and 12th weeks | up to 12th week
  The Cervical Radiculopathy Impact Scale (CRIS) is developed a self-report questionnaire which covers the measurement of symptoms and limitations in patients with cervical radiculopathy due to irradiating pain, tingling sensations and sensory loss in the arm in combination with neck disability. It is divided into 3 subgroups as symptoms, energy&posture and activities &actions consist of 21 items. Every subgroup of the questionnaire has a score scale between 0 and 100 Each question measures from 0 to 5 is calculated. Higher scores mean worse outcome.
Change from baseline Pain detect questionnaire (PD-Q) at 4th and 12th weeks | up to 12th week
  It's used to detect neuropathic pain components in chronic neck pain. It contains 2 items related to the spatial and temporal characteristics of the pain pattern and 7 sensory descriptive items. Minimum 0 and maximum of 38 points can be obtained. Higher scores mean worse outcome. PD-Q cut-off scores are ≤ 12 (a neuropathic component is unlikely) and ≥ 19 (a neuropathic component is likely).

CONTACTS AND LOCATIONS:
Overall Officials: Songül İNCE, MD, Principal Investigator — Afyonkarahisar Health Sciences University; Nuran EYVAZ, MD, Principal Investigator — Afyonkarahisar Health Sciences University
Locations (1):
- AFYON, Afyonkarahisar, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Konstantinovic LM, Cutovic MR, Milovanovic AN, Jovic SJ, Dragin AS, Letic MDj, Miler VM. Low-level laser therapy for acute neck pain with radiculopathy: a double-blind placebo-controlled randomized study. Pain Med. 2010 Aug;11(8):1169-78. doi: 10.1111/j.1526-4637.2010.00907.x. PMID 20704667
- [Background] Song HJ, Seo HJ, Lee Y, Kim SK. Effectiveness of high-intensity laser therapy in the treatment of musculoskeletal disorders: A systematic review and meta-analysis of randomized controlled trials. Medicine (Baltimore). 2018 Dec;97(51):e13126. doi: 10.1097/MD.0000000000013126. PMID 30572425
- [Background] Alayat MS, Mohamed AA, Helal OF, Khaled OA. Efficacy of high-intensity laser therapy in the treatment of chronic neck pain: a randomized double-blind placebo-control trial. Lasers Med Sci. 2016 May;31(4):687-94. doi: 10.1007/s10103-016-1910-2. Epub 2016 Feb 25. PMID 26914684